CLINICAL TRIAL: NCT00677625
Title: Pediatric Liver Disease and Liver Transplant Database
Brief Title: Pediatric Liver Database
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Grzegorz Telega, Associate Professor of Pediatrics, Medical College of Wisconsin
Other Study IDs: CHW 03/64 HRRC 188-03
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Liver Disease; Liver Transplant
Keywords: Liver; Transplant
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver Disease (LD): These child subjects have some form of liver disease (including those who need a liver transplant) or have already had a liver transplant.

SUMMARY:
The purpose of this study is to collect data to examine and characterize the clinical outcomes of pediatric patients diagnosed with any liver disease at Children's Hospital of Wisconsin.

DETAILED DESCRIPTION:
In this study, medical information which is routinely obtained on children with any liver diseases, or children who have had a liver transplant will be entered into a database. No extra tests are done for participating in this study, and no extra visits to the doctor are required. The clinical data collected is then entered into a database and followed longitudinally. The information obtained from this study will help researchers learn more about pediatric liver disease, therefore providing better routine clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age
* newly diagnosed with a liver disease, currently listed for liver transplant, or who are being considered for liver transplantation and evaluated
* receive a liver transplant prior to their eighteenth birthday

Exclusion Criteria:

* Patients decline participation.
* Patients have no liver diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All child subjects will be recruited from the Hepatology Clinic at Children's Hospital of Wisconsin
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2003-06; Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Telega, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States